CLINICAL TRIAL: NCT04210544
Title: Effect of a Protein Intake on the Feeling of Hunger / Satiety in Men and Women Through an Acute Postprandial Study
Brief Title: Protein Intake and Satiety: a Postprandial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Marian Zulet, Professor, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.069
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Satiety
Keywords: Satiety; Hunger; Obesity; Ghrelin; Visual Analogue Scale; Gastrointestinal hormones; Energy compensation
MeSH Terms: conditions — Obesity | interventions — Caseins; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary protein (Experimental): Postprandial effects after consuming 20 g of a experimental dietary protein mixed with 250 g of custard and to drink of 50 mL of water served in a glass.
  Interventions: Dietary Supplement: Experimental dietary protein
- Casein (Active Comparator): Postprandial effects after consuming 20 g of casein mixed with 250 g of custard and to drink of 50 mL of water served in a glass.
  Interventions: Dietary Supplement: Casein
- Water (Placebo Comparator): Postprandial effects after consuming 20 g of water mixed with 250 g of custard and to drink of 50 mL of water served in a glass.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Experimental dietary protein — Breakfast intake consisted on a 250 g custard intake mixed with 20 g of the experimental protein accompanied by a glass with 50 mL water.
  Arms: Dietary protein
Dietary Supplement: Casein — Breakfast intake consisted on a 250 g custard intake mixed with 20 g of casein accompanied by a glass with 50 mL water.
  Arms: Casein
Dietary Supplement: Water — Breakfast intake consisted on a 250 g custard intake mixed with 20 g of water accompanied by a glass with 50 mL water.
  Arms: Water

SUMMARY:
Obesity is considered the emerging epidemic of the 21st century, becoming one of the major public health problems. Excessive body weight increases morbidity and mortality risk, while decreases the quality of life and expectance. The prevalence of obesity almost has doubled in the last 20 years. According to the World Health Organization, 39% of the population is overweight and 13% of the population is obese.

Obesity is a multifactorial origin disease, where genetic plays an important role. However, lifestyle factors, such as unhealthy diets and physical inactivity are the main cause for the development of obesity and associated comorbidities such as hypertension, dyslipidemia, diabetes and even some types of cancer. The prevention and control of obesity as well as its comorbidities requires interventions at individual and population level.

Intervention studies based on hypocaloric diets show poor adherence in the long term. Moreover, high energy density diets accompanied by snacking between meals contribute to weight gain. Therefore, the inclusion of bioactive compounds with satiating capacity within healthy and personalized dietary patterns could be a strategy to improve adherence in a dietary plan, and consequently reduce morbidity and mortality rates associated to obesity.

Considering this background, the general aim of this investigation is to perform an acute postprandial study to evaluate the effect of a dietary protein intake on the feeling of hunger and satiety. To carry out this objective, different data will be analysed, such as the measurement of gut hormone circulating concentrations, lipid and glucose profile, energy compensation after the postprandial period and the total energy intake during the day.

DETAILED DESCRIPTION:
This study is designed as a crossover, randomized, three-arm postprandial study. All participants attend the Nutrition Intervention Unit of the Centre for Nutrition Research in the University of Navarra three times separated by at least one week. The day before each study day, participants should avoid vigorous physical exercise, alcohol consumption or high-fiber food consumption. Moreover, they are asked to follow a standardized dinner before 9 pm.

On each study day, participants visit the Nutrition Intervention Unit in fasting state. After 5 minutes rest and having answered the first hunger / satiety visual analogue scale (VAS) questionnaire, blood pressure is measured. After that, participant are asked to collect a baseline urine sample.

Once the cannulation is placed, first blood collection is performed in fasting state (time 0). Then, the participant is provided with the randomly assigned standardized breakfast (250 g of custard) with the addition of 20 g of experimental protein or 20 g of casein or 20 g of water. After custard consumption, volunteer is asked to drink 50 mL of water.

When participant finishes the breakfast, the time is registered and every 15 minutes the participant have to complete a VAS questionnaire (15´, 30´, 45´, 60´, 75´ and 90´). Moreover, blood samples are drawn at different time points after breakfast intake (15´, 30´, 60´ and 90´). The cannula is removed when the last blood sample is collected. In addition, participants are asked to collect the urine sample at 90 minutes postingestion and to fill a questionnaire about gastrointestinal symptoms.

Finally, participant is offered an ad libitum lunch (ham and cheese sandwiches) to eat until feeling comfortably satiated. Once completed, participant leaves the Centre for Nutrition Research with the necessary material to register the food intake (solids and liquids) during the rest of the day. Likewise, the participant is provided with the questionnaire of gastrointestinal symptoms to be filled before the dinner of the same day.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 20-65 years.
* Overweight or obese (BMI: 24.9 - 34.9 kg / m2).
* Physical characteristics and vital signs normal or clinically without relevance to the experiment.
* Volunteers undergoing drug treatment will be included if the dose is stable for at least three months before the start of the study with the exception of treatments that alter gastrointestinal function, lipid lowering and antidiabetics treatments.
* Able to understand and be willing to sign the informed consent form and to follow all the study procedures and requirements.

Exclusion Criteria:

* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasia, active peptic ulcers, chronic inflammatory diseases or malabsorption.
* Consuming more than 14 units of alcohol intake per week in women, or more than 21 units per week in men.
* Pregnancy or lactation.
* Subjects who have undergone surgical interventions with permanent sequelae (for example, gastroduodenostomy).
* Subjects with some liver disease.
* Subjects with some type of cancer or in treatment of it, or less than 5 years after its eradication.
* Subjects with allergy to any component of the products under study or some other food that interferes and makes difficult to follow the study.
* Subjects that present some kind of cognitive and / or psychical impairment.
* Subjects with poor collaboration, or with difficulty to follow the study procedures.
* Subjects who exhibit restrictive or specific behaviors in the diet (Eating Attitude Test-26 equal or more than 20 points).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Baseline subjective hunger | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm, for the quantification the perceived hunger before the experimental custard intake.
Postprandial subjective hunger | Up to 90 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived hunger measured at 15, 30, 45, 60, 75 and 90 minutes after experimental custard intake.
Baseline subjective fullness | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived fullness before experimental custard intake.
Postprandial subjective fullness | Up to 90 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived hunger measured at 15, 30, 45, 60, 75 and 90 minutes after experimental custard intake.
Baseline subjective satiety | Baseline
  Visual analogue scale rating in a scale from 0 to100 mm for the quantification of the perceived fullness before experimental custard intake.
Postprandial subjective satiety | Up to 90 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived hunger measured at 15, 30, 45, 60, 75 and 90 minutes after experimental custard intake.
Baseline subjective desire to eat | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived fullness before experimental custard intake at baseline.
Postprandial subjective desire to eat | Up to 90 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived hunger measured at 15, 30, 45, 60, 75 and 90 minutes after experimental custard intake.
Baseline subjective thirst | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived fullness before experimental custard intake.
Postprandial subjective thirst | Up to 90 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived hunger measured at 15, 30, 45, 60, 75 and 90 minutes after experimental custard intake.
Baseline blood ghrelin concentration | Baseline
  Blood ghrelin concentration before experimental custard intake.
Postprandial blood ghrelin concentration | Up to 90 minutes
  Blood ghrelin concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Ad libitum food intake | 90 minutes
  Quantification of food intake after the 90 minutes of postprandial period.

SECONDARY OUTCOMES:
Baseline weight | Baseline
  Baseline weight of participants will be reported in kg and will be performed in the first visit.
Baseline height | Baseline
  Baseline height of participants will be reported in cm and will be performed in the first visit.
Baseline body mass index | Baseline
  To calculate baseline body mass index weight and height will be combined to report BMI in kg/m^2
Baseline waist circumference | Baseline
  Baseline waist circumference will be reported in cm and will be performed in the first visit
Baseline systolic blood pressure | Baseline
  Baseline systolic blood pressure will be reported in mmHg at each visit
Baseline diastolic blood pressure | Baseline
  Baseline diastolic blood pressure will be reported in mmHg at each visit
Baseline heart rate | Baseline
  Baseline heart rate will be reported in beat/minute at each visit
Baseline blood glucose concentration | Baseline
  Blood glucose levels before experimental custard intake
Postprandial blood glucose concentration | Up to 90 minutes
  Blood glucose measured at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood insulin concentration | Baseline
  Blood insulin levels before experimental custard intake
Postprandial blood insulin concentration | Up to 90 minutes
  Blood insulin measured at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline insulin resistance index (HOMA) | Baseline
  Insulin resistance index (HOMA) before experimental custard intake
Postprandial insulin resistance index (HOMA) | Up to 90 minutes
  Insulin resistance index (HOMA) at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood total cholesterol concentration | Baseline
  Blood total cholesterol concentration before experimental custard intake
Postprandial blood total cholesterol concentration | Up to 90 minutes
  Blood total cholesterol concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood high density lipoprotein cholesterol (HDL) concentration | Baseline
  Blood high density lipoprotein cholesterol (HDL) concentration before experimental custard intake
Postprandial blood high density lipoprotein cholesterol (HDL) concentration | Up to 90 minutes
  Blood high density lipoprotein cholesterol (HDL) concentration at 15, 30, 60 and 90 minutes after consuming 250 g of the experimental custard.
Baseline blood low density lipoprotein cholesterol (LDL) concentration | Baseline
  Blood low density lipoprotein cholesterol (LDL) concentration before experimental custard intake
Postprandial blood low density lipoprotein cholesterol (LDL) cholesterol concentration | Up to 90 minutes
  Low density lipoprotein cholesterol (LDL) concentration at 15, 30, 60 and 90 minutes after experimental custard intake
Baseline blood triglyceride concentration | Baseline
  Blood triglyceride concentration before experimental custard intake
Postprandial blood triglyceride concentration | Up to 90 minutes
  Blood triglyceride concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood cholecystokinin (CCK) concentration | Baseline
  Blood cholecystokinin (CCK) concentration before experimental custard intake
Postprandial blood cholecystokinin (CCK) concentration | Up to 90 minutes
  Blood cholecystokinin (CCK) concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood glucagon like peptide-1 concentration | Baseline
  Blood glucagon like peptide-1 concentration concentration before experimental custard intake
Postprandial blood glucagon like peptide-1 concentration | Up to 90 minutes
  Blood glucagon like peptide-1 concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood peptide YY (PYY) concentration | Baseline
  Blood peptide YY (PYY) concentration before experimental custard intake
Postprandial blood peptide YY (PYY) concentration | Up to 90 minutes
  Blood peptide YY (PYY) concentration at 15, 30, 60 and 90 minutes after experimental
Questionnaire about gastrointestinal symptoms (1) | 90 minutes
  Gastrointestinal questionnaire at 90 minutes of consuming the experimental custard.
Questionnaire about gastrointestinal symptoms (2) | Before dinner of the experimental day
  Gastrointestinal questionnaire before dinner of the experimental day.
Quantification of food intake during the rest of the day | During the whole day of the experimental day.
  Food record calibration from the end of the ad libitum lunch until go to sleep.
Baseline blood apolipoprotein concentration | Baseline
  Blood apolipoproteins concentration before experimental custard intake
Postprandial blood apolipoprotein concentration | Up to 90 minutes
  Blood apolipoprotein concentration at 15, 30, 60 and 90 minutes after experimental custard intake.
Baseline blood concentration of reference amino acid of the experimental protein. | Baseline
  Baseline blood concentration of reference amino acids of the experimental protein.
Postprandial blood concentration of reference amino acid of the experimental protein | Up to 90 minutes
  Blood concentration (15, 30, 60 and 90 minutes) of reference amino acid of the experimental protein after the experimental custard intake.
Baseline urine concentration of reference amino acid of the experimental protein. | Baseline
  Baseline urine concentration of reference amino acid of the experimental protein.
Urine concentration of reference amino acid of the experimental protein at 90 minutes post ingestion | 90 minutes
  Urine concentration of reference amino acid of the experimental protein at 90 minutes post ingestion

CONTACTS AND LOCATIONS:
Overall Officials: M Ángeles Zulet Alzórriz, Professor, Principal Investigator — Centre for Nutrition Research - University of Navarra
Locations (1):
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No